Effects of the COVID-19 Health Emergency on the Biopsychosocial Health of Rural Residents of New Mexico using Mixed Methods

IRB: 20-266

NCT04409535

Document Date: May 6, 2020

Effects of the COVID-19 Health Emergency on the Biopsychosocial Health of Rural Residents of New Mexico using Mixed Methods

IRB: 20-266

**Principal Investigator:** 

Carla Wilhite, Assistant Professor, Dept. of Peds, HSSB Room 140, 272-3324, cwilhite@salud.unm.edu

Name, Title, Department, Building, Phone, Fax, E-mail address

4. Co-Investigators and key personnel:

Janet L. Poole, Professor, Dept. of Peds, HSSB Room 140, 277-1753, <a href="mailto:ilpoole@salud.unm.edu">ilpoole@salud.unm.edu</a> Timothy Dionne, Assistant Professor, HSSB Room 140, 27701753, tdionne@salud.unm.edu

DATA ANALYSIS PLAN

Qualitative

Per the procedures in Creswell data analysis of the interviews was planned as a multi-step process. The data analysis was tasked to the experts at the UNM-Center for Translational Research (CTSC) using NVivo software. First, the data was organized and prepared for analysis. The interviews were transcribed, and auditory confirmation of the transcript was conducted by the researcher. All the electronic data was sorted into the corresponding file allocated for the participant, sans identifiers, for purposes of backup. The information was secured by the CTSC.

Using the recommendations of Creswell for analyzing phenomenology, the data was scanned to gain a general sense of what each participant was saying about the phenomenon of the COVID experience. Further coding of the data was conducted to develop nascent themes or nodes. Thematic analysis was carried out by the CTSC and verified with the researchers. Every effort was made to ensure the trustworthiness of the report and the analysis also subjected to peer debriefing and an independent auditor verified the findings.

Quantitative:

Quantitative analysis of the WHOQOL-BREF was conducted by Dr. Timothy Dionne with the assistance of a statistician from the CTSC and a graduate student.